CLINICAL TRIAL: NCT00889499
Title: Modulation of Central Hypersensitivity in Chronic Musculoskeletal Pain by Intravenous Tropisetron
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Michele Curatolo / Prof., Inselspital, Bern University Hospital, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KEK 146/04
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Pain; Chronic Disease
MeSH Terms: conditions — Pain; Chronic Disease | interventions — Tropisetron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Crossover study (Placebo Comparator): Crossover study
  Interventions: Drug: Tropisetron 2 mg
- 2 (Placebo Comparator): Crossover Study
  Interventions: Drug: Tropisetron 5mg
- 3 (Placebo Comparator): Crossover Study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tropisetron 2 mg — Antagonist of the 5HT3 receptor.
  Arms: Crossover study
Drug: Tropisetron 5mg — Antagonist of the 5HT3 receptor.
  Arms: 2
Drug: Placebo — NHCL 0,9%
  Arms: 3

SUMMARY:
Chronic pain is associated with hypersensitivity of the central nervous system. The drug under investigation (tropisetron) has been shown in animal studies to attenuate central hypersensitivity. It has therefore the potential to be effective in chronic pain. We compare two doses of tropisetron with placebo in patients with chronic pain. We measure pain intensity and parameters that assess central hypersensitivity.

DETAILED DESCRIPTION:
Background

Prolonged afferent nociceptive input induces an increase in the excitability of central sensory neurons. The hyperexcitable neurons amplify the nociceptive signal, thereby producing an exaggerated pain response. This state of central hypersensitivity very likely contributes to pain and disability in patients, even in the presence of limited tissue damage.

The 5-hydroxytryptamine-3 (5-HT-3) receptor is involved in spinal nociceptive transmission. After experimentally induced inflammation, the selective 5-HT-3 receptor antagonist ondansetron inhibited the electrically evoked responses of dorsal horn neurones, but had no effect on these responses in the absence of inflammation. Importantly, the origin of this pathway is a spino-brainstem-spinal loop that includes areas of the brain involved in emotional and affective responses to pain. This suggests that the 5-HT-3 receptors have no significant role under normal conditions, but are activated by peripheral inflammation and contribute to spinal cord hyperexcitability. Their activity could be driven by anxiety and fear.

Spinal cord hyperexcitability elicited by trauma, inflammation or surgery is influenced by descending facilitatory and inhibitory pathways. The periaqueductal grey and endogenous opioid peptides play a central role in the inhibition of spinal cord neuronal responses. Release of enkephalin at supraspinal and spinal levels is evoked by noxious stimulation. Further inhibitory modulation is exerted by serotonergic and noradrenergic systems. These mechanisms may underlie a possible role of psychological disturbances in the spinal cord processing of nociceptive and non-nociceptive stimuli.

While central hypersensitivity mechanisms have been extensively investigated in the animal, data in patients are sparse. In patients, direct measurements at spinal cord or brain neurons can not be made. Therefore, it is impossible to provide direct evidence for neuronal hyperexcitability. However, hypersensitivity can be investigated indirectly by quantitative sensory tests. Typically, hypersensitivity is detected when sensory stimulation evokes pain at stimulus intensities that do not induce pain in normal subjects (lower pain threshold) or when a standardised painful stimulus evokes stronger pain in patients than in normal subjects. Other methods to explore the sensory system are available, but a detailed description is beyond the scope of this section. Whenever pain hypersensitivity is observed after sensory stimulation of healthy areas, its cause must be a hyperexcitability of the central nervous system. Indeed, there is no evidence that peripheral mechanisms could account for a higher pain sensitivity at healthy tissues.

Using the sensory tests, central hyperexcitability has been detected in different chronic musculoskeletal pain syndromes, such as neck pain after whiplash injury, fibromyalgia, osteoarthritis and temporomandibular disorders. Objective electrophysiological evidence for spinal cord hypersensitivity has recently been provided for patients with neck pain after whiplash injury and in fibromyalgia patients.

Few attempts have been made to modulate central hypersensitivity in patients. Infiltration of the local anaesthetic into the painful and tender muscles of patients with chronic neck pain did not reduce either neck pain nor pain thresholds. This indicated that the source of pain was not located in the infiltrated muscles and central hypersensitivity was not maintained by a nociceptive input arising from these muscles, at least in the patient population investigated. Selective 5-HT-3 receptor antagonists have proven effective in patients with fibromyalgia. Because fibromyalgia is associated with central hypersensitivity, one can postulate an activation of the spinal 5-HT-3 system as one of the mechanisms involved in the pathophysiology of this pain syndrome. The facilitatory pathway mediated by this receptor involves parts of the brain associated with emotional and affective responses to pain. An effect of selective 5-HT-3 receptor antagonists on other musculoskeletal pain syndromes associated with central hypersensitivity, such as whiplash or osteoarthritis, can not be ruled out. In a recent placebo-controlled study, a single intravenous injection of the selective 5-HT-3 receptor antagonist Ondansetron produced pain relief in patients with neuropathic pain.

Objective

The project will address the following main hypotheses. A. Reduction in pain and central hypersensitivity is accomplished by administration of the 5-HT-3 antagonist tropisetron.

B. The analgesic effect of Tropisetron is predicted in individual patients by the electrophysiological measurements that assess central hypersensitivity.

Methods

Pain intensity is assessed by the visual analogue scale (VAS). The following measures of central hypersensitivity will be employed: pain detection and pain tolerance threshold to electrical stimulation, heat and cold stimulation, spinal nociceptive reflexes, assessment of reflex receptive fields and temporal summation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain
* Pain duration at least 6 months

Exclusion Criteria:

* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Pain intensity (VAS score) | 2 h

SECONDARY OUTCOMES:
Measures of central hypersensitivity | 2 h

CONTACTS AND LOCATIONS:
Overall Officials: Michele Curatolo, Prof, Study Director — Inselspital, Bern University Hospital
Locations (1):
- Dep. of Anesthesiology and Pain Therapy, Bern University Hospital, Inselspital, Bern, Switzerland